CLINICAL TRIAL: NCT03595852
Title: Preoperative Antibiotic Prophylaxis Versus Placebo in Clean, Non-prosthetic Surgery at CHUK. Impact on Surgical Site Infections and Patient Cost.
Brief Title: Antibiotic Prophylaxis in Clean Surgery. Impact on Surgical Site Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Responsible Party: Principal Investigator, Isaie Sibomana, Resident in surgery, University of Rwanda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1234
Record Dates: First submitted 2017-08-03; First posted 2018-07-23 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: antibiotic prophylaxis versus placebo in clean non prosthetic surgery. impact on surgical site infection and patient cost.
Who Masked: Participant, Investigator
Masking Description: patients and investigator will be blinded for intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylaxis (Experimental): The intervention will be a single dose of prophylactic antibiotic (cefazolin): 2 gr in adults or 3 gr for patients weighing >120Kg or 30mg/kg in children given within 30-60 minutes prior to skin incision.
  Interventions: Drug: Cefazolin
- No prophylaxis (Placebo Comparator): The control group will receive a similarly looking prepared placebo injection (normal saline placebos for injection) 30-60 minutes prior to incision.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Cefazolin — Cefazolin will be given to patients in the experimental arm prophylactically prior to surgery
  Other Names: ancef
  Arms: Prophylaxis
Drug: Placebos — IV normal saline will be given to patients 30-60 minutes prior to incision
  Other Names: saline
  Arms: No prophylaxis

SUMMARY:
This is a randomized control study of antibiotic uses in clean non prosthetic surgeries. One group will be given antibiotic prophylaxis, other will receive a placebo. The primary outcome will be the rate of surgical site infection in 2 groups.

DETAILED DESCRIPTION:
I will conduct a randomized controlled trial (RCT) of antibiotic prophylaxis versus placebo in clean, non-prosthetic, elective procedures. The intervention will be a single dose of prophylactic antibiotic (cefazolin): 2 gr in adults or 3 gr for patients weighing >120Kg and 30mg/kg in children) within 30-60 minutes prior to skin incision. The control group will receive a similarly prepared placebo injection (water for injection) 30-60 minutes prior to incision.

I will randomize patients in a 1:1 allocation ratio using a simple randomization. Patients will randomly pick an envelope with a number allocating to antibiotic prophylaxis or placebo. Patients and caretakers will be blinded to the intervention. The surgeon will also be blinded to the intervention. The antibiotic (or placebo) will be pre-mixed by the study investigator and administered by the anesthetist.

Other preventive measures for surgical site infection (SSIs) such as effective surgical hand scrub, proper skin preparation with povidone and sterility of materials and instrument will be applied systematically in all groups. Dressing of the wound will be removed 48 hours after operation and no further dressing will be required. Patients will be followed for development of SSI documented by surgeon at discharge and will be called after 30 days of surgery to address any sign of SSI.

ELIGIBILITY:
Inclusion Criteria:

* - All elective non-prosthetic surgical procedures such as hernia, thyroid, hydrocele, undescended testes surgery, removal of orthopedic implants, low risk breast surgical procedures and other all procedures deemed to be clean.

Exclusion Criteria:

* - Emergency cases
* Any patient with American Society of Anesthesiologists Score (ASA)>2
* Procedures lasting more than 2 hours
* Patients who were taking antibiotics 2 days prior to operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days post operative
  surgical wounds will be accessed for signs of surgical site infection at discharge by a treating surgeon and patients will be called 30 days after operation for signs of surgical site infection

SECONDARY OUTCOMES:
mortality | 48 hours post operation
  death
morbidity | 48 hours post operation
  morbidity will be defined as any one of the following clinical diagnoses made by a treating surgeon: unplanned reoperation, healthcare associated infection, pneumonia, cardiac arrest, pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: FAUSTIN NTIRENGANYA, MMed, FCS, Study Director — fostino21@yahoo.fr
Locations (1):
- Kigali University Teaching Hospital (Chuk), Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD to other researchers